CLINICAL TRIAL: NCT06587035
Title: A Multicenter, Non-interventional Prospective Active Surveillance Study Among Participants Receiving Somatrogon Under Routine Clinical Care in India
Brief Title: A Study to Learn About Somatrogon in Patients With Pediatric Growth Hormone Deficiency (p GHD) in India.
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C0311026; NCT06587035 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Dwarfism, Pituitary
Keywords: Somatrogon, Safety
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somatrogon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients of pediatric growth hormone deficiency
  Interventions: Drug: Somatrogon

INTERVENTIONS:
Drug: Somatrogon — Long-acting growth hormone for pediatric growth hormone deficiency.

SUMMARY:
The purpose of this study is to learn about the safety of Somatrogon for the treatment of pediatric growth hormone deficiency (p GHD) in India.

Pediatric GHD is a condition caused by too less amounts of growth hormone in the body. Children with GHD have a short height. GHD can be present at birth or develop later. The condition occurs if the pituitary gland makes too little growth hormone. This is a small gland at the bottom of the brain that releases hormones that affect growth and other body functions.

This study is seeking for participants who are:

* confirmed with p GHD.
* given Somatrogon to be taken as an injection.

The safety of Somatrogon injection will be checked based on side effects. These side effects can happen within 3 years after taking Somatrogon. A side effect is something (expected or unexpected) that you feel was caused by a medicine or treatment you take. The study doctor will collect side effect information and put the information on patient's case form.

Follow-up of the patient's will be performed via clinic re-visit or over a call. It is not a rule for the participants to visit the clinic in this study.

This study will help to see if Somatrogon is safe.

ELIGIBILITY:
Inclusion Criteria:

* Prescription of Somatrogon for p GHD in participants aged 3 years or more.
* Evidence of a personally signed and dated informed consent document indicating that the participant (or a legally acceptable representative) has been informed and agree to all pertinent aspects of the study. Assent will also be sought from children of applicable age in line with national guidance. In all cases, the treating physician responsible for enrolling the participant into the study will assess the appropriateness of gaining assent from a participant (or a legally acceptable representative) at their discretion during routine clinical care.

Exclusion Criteria:

* Participation in any interventional clinical trials at the time of enrollment.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants treated with Somatrogon will be followed by the treating physician as per routine clinical practice, who will collect and enter relevant participant data onto case report forms (CRFs).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2028-09-05 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events in participants on Somatrogon | 3 years

SECONDARY OUTCOMES:
Number of participants reporting missed injections with Somatrogon in order to evaluate treatment adherence | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- India (4):
  - Shivajoyti Clinic, Bengaluru, Karnataka
  - Apollo Children's Hospital, Chennai, Tamil Nadu
  - G Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
  - Apollo Speciality Hospital, Madurai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0311026